CLINICAL TRIAL: NCT07300592
Title: Development of a Static Balance Assessment Tool for High-Functioning Older Adults
Brief Title: Development of a Static Balance Assessment Tool for High-Functioning Older Adults (KSVGH25-CT3-09)
Acronym: KSVGH25-CT3-09
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jia-Ling Hong (Other)
Responsible Party: Sponsor-Investigator, Jia-Ling Hong, Kaohsiung Municipal United Hospital, Kaohsiung Municipal United Hospital
Organization: Kaohsiung Municipal United Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KSVGH25-CT3-09
Record Dates: First submitted 2025-11-22; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Balance Assessment; Postural Balance; Older Adults, Balance
Keywords: Static balance assessment

STUDY DESIGN:
Intervention Model Description: All participants will receive the same assessment procedures, including body composition measurement, open-eyes/closed-eyes single-leg stance, and the Balance Error Scoring System under firm and foam surface conditions. Two identical assessment sessions will be conducted 5-7 days apart to evaluate test-retest reliability.
Masking Description: Outcome assessors who review video recordings will be blinded to the on-site assessment results to reduce scoring bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Static Balance Assessment Group (Experimental): Participants will undergo body composition measurement, open-eyes and closed-eyes single-leg stance test, and Balance Error Scoring System testing under firm and foam surface conditions. Each participant will complete two identical sessions, 5-7 days apart, with both on-site scoring and video-based scoring to determine test-retest reliability.
  Interventions: Other: Static Balance Assessment Protocol

INTERVENTIONS:
Other: Static Balance Assessment Protocol — Participants will undergo a standardized static balance assessment protocol, including open-eyes and closed-eyes single-leg stance tests, as well as Balance Error Scoring System (BESS) testing under firm and foam surface conditions. Each participant will complete two identical sessions, 5-7 days apart, with both on-site scoring and video-based scoring performed by trained assessors to determine test-retest reliability.

SUMMARY:
This single-center interventional study aims to develop and validate a static balance assessment tool tailored for high-functioning older adults. Participants aged 65 years or older, who achieve a perfect score on the Short Physical Performance Battery and can maintain an open-eyes single-leg stance for at least 10 seconds, will be recruited. The assessment includes body composition measurement, open-eyes/closed-eyes single-leg stance, and the Balance Error Scoring System under firm and foam surface conditions. Each participant will undergo two testing sessions, 5-7 days apart, with both on-site and video-based scoring to determine test-retest reliability. The expected outcome is the development of an accurate and highly applicable static balance measurement tool to support healthy aging and fall prevention in community and long-term care settings.

DETAILED DESCRIPTION:
The study is conducted at Kaohsiung Municipal United Hospital, Taiwan, with the objective of creating a static balance assessment tool specifically designed for older adults who are physically high-functioning. Traditional balance tests, such as the open-eyes single-leg stance with a 30-second limit, often produce ceiling effects in this population, making it difficult to detect subtle differences in balance ability or evaluate the benefits of exercise programs. To address this limitation, the current study extends the open-eyes single-leg stance to a maximum of 60 seconds and incorporates a closed-eyes condition to increase task difficulty.

In addition, the Balance Error Scoring System, originally developed for concussion assessment, will be adapted for older adults. Balance Error Scoring System testing will be conducted under six conditions: double-leg stance, tandem stance, and single-leg stance, each performed on both firm and foam surfaces with eyes closed. This design simulates balance challenges encountered in daily life while minimizing fall risk.

Eligible participants (n=50) will be community-dwelling older adults aged ≥65 years, with perfect Short Physical Performance Battery scores and no recent lower limb injuries or neurological conditions. Each participant will complete two identical assessment sessions, spaced 5-7 days apart. Both on-site evaluators and independent assessors reviewing video recordings will score performance. The primary outcome is the test-retest reliability of each balance measure, quantified through statistical analysis.

The anticipated benefit of this study is to establish a reliable, sensitive, and practical balance assessment protocol that can be implemented in community health programs, long-term care facilities, and research settings. This tool aims to improve early detection of balance decline, guide intervention planning, and ultimately contribute to fall prevention and healthy aging initiatives in aging societies.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 85 years
* Able to walk independently without assistive devices
* No self-reported balance disorders or history of recurrent falls in the past 6 months
* Cognitively intact (Mini-Mental State Examination score ≥ 24)
* Willing and able to provide informed consent

Exclusion Criteria:

* Diagnosed neurological disorders affecting balance (e.g., Parkinson's disease, stroke with residual deficits)
* Diagnosed neurological disorders affecting balance (e.g., Parkinson's disease, stroke with residual deficits)
* Severe visual or vestibular impairment uncorrected by aids
* Lower limb musculoskeletal disorders that limit mobility
* Current participation in other interventional clinical trials
* Unstable cardiovascular conditions (e.g., uncontrolled hypertension, recent myocardial infarction)
* Severe visual or vestibular impairment uncorrected by aids
* Lower limb musculoskeletal disorders that limit mobility
* Current participation in other interventional clinical trials
* Unstable cardiovascular conditions (e.g., uncontrolled hypertension, recent myocardial infarction)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Test-Retest Reliability of Static Balance Assessment Scores | Within 7 days after the first assessment
  Description: Reliability will be evaluated using intra-class correlation coefficient (ICC) and Spearman correlation coefficient (ρ) between session 1 and session 2 scores for the following static balance tests:
  Single-leg stance with eyes open Single-leg stance with eyes closed Balance Error Scoring System (BESS) under various surface conditions Scale Name: Balance Error Scoring System (BESS) Score Range: 0 (best balance) to 60 (worst balance) Interpretation: Higher BESS scores indicate worse balance performance.
Short Physical Performance Battery (SPPB) - 4-Meter Walk Test | Within 7 days after the first assessment
  Unit of Measure: Seconds (s) Description: Measures usual gait speed over a 4-meter distance. Interpretation: Lower time indicates better performance.
Short Physical Performance Battery (SPPB) - 5-Times Sit-to-Stand Test | Within 7 days after the first assessment
  Unit of Measure: Seconds (s) Description: Measures lower-limb strength and functional mobility. Interpretation: Lower time indicates better performance.

SECONDARY OUTCOMES:
Body Height | At baseline (first assessment)
  Unit of Measure: Centimeters (cm)
Body Weight | At baseline (first assessment)
  Unit of Measure: Kilograms (kg)
Body Mass Index (BMI) | At baseline (first assessment)
  Unit of Measure: Kilograms per square meter (kg/m²) Calculated as weight in kilograms divided by height in meters squared.
Whole-Body Skeletal Muscle Mass | At baseline (first assessment)
  Unit of Measure: Kilograms (kg)
  Description:
  Whole-body skeletal muscle mass will be measured using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer. Participants will stand barefoot and hold hand electrodes during the assessment.
Single-Leg Stance Test - Eyes Open | Within 7 days after the first assessment
  Test Name: Single-Leg Stance Test (Eyes Open) Unit of Measure: Seconds (s) Description: Participant stands unassisted on one leg with eyes open. The time is recorded until balance is lost or foot touches the ground.
  Interpretation: Longer time indicates better static balance performance.
Single-Leg Stance Test - Eyes Closed | Within 7 days after the first assessment
  Test Name: Single-Leg Stance Test (Eyes Closed) Unit of Measure: Seconds (s) Description: Participant stands unassisted on one leg with eyes closed. The time is recorded until balance is lost or foot touches the ground.
  Interpretation: Longer time indicates better static balance performance.
Whole-Body Muscle Mass | At baseline (first assessment)
  Unit of Measure: Kilograms (kg)
  Description:
  Whole-body muscle mass will be assessed using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.
Segmental Muscle Mass - Upper and Lower Limbs and Trunk | At baseline (first assessment)
  Unit of Measure: Kilograms (kg)
  Description:
  Segmental muscle mass of the right upper limb, left upper limb, trunk, right lower limb, and left lower limb will be measured using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.
Whole-Body Body Fat Percentage | At baseline (first assessment)
  Unit of Measure: Percentage (%)
  Description:
  Whole-body body fat percentage will be measured using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.
Segmental Body Fat Percentage | At baseline (first assessment)
  Unit of Measure: Percentage (%)
  Description:
  Segmental body fat percentage of the right upper limb, left upper limb, trunk, right lower limb, and left lower limb will be measured using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.
Visceral Fat Level | At baseline (first assessment)
  Unit of Measure: Arbitrary units (BIA-derived level)
  Description:
  Visceral fat level will be estimated using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.
Basal Metabolic Rate | At baseline (first assessment)
  Unit of Measure: Kilocalories per day (kcal/day)
  Description:
  Basal metabolic rate will be estimated using bioelectrical impedance analysis (BIA) with the TANITA BC-545N body composition analyzer.

OTHER OUTCOMES:
Fall Frequency | At baseline (first assessment)
  Unit: Number of falls in past 12 months
Living Status | At baseline (first assessment)
  Unit: Categorical (living alone / with others)
Education Level | At baseline (first assessment)
  Unit: Categorical (elementary, high school, etc.)
Exercise Habit | At baseline (first assessment)
  Unit: Categorical (Yes / No)
Exercise Duration | At baseline (first assessment)
  Unit: Hours per week (hr/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Municipal United Hospital, Kaohsiung City, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. The decision is based on institutional policy and the need to protect participant privacy and confidentiality. Only aggregated results will be reported in publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT07300592/Prot_SAP_000.pdf